CLINICAL TRIAL: NCT06412653
Title: Prospective Pilot Trial to Address the Feasibility and Safety of Treatment With Oral Zinc in GNAO1 Associated Disorders
Brief Title: Prospective Pilot Trial to Address Feasibility and Safety of Oral Zinc in GNAO1 Associated Disorders
Acronym: ZINCGNAO1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's University Hospital Cologne, Germany (Other)
Collaborators: The Clinical Trials Centre Cologne (Other); University of Cologne (Other); University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Moritz Thiel, MD, Pediatrician in pediatric neurology, Children's University Hospital Cologne, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-5275
Record Dates: First submitted 2024-02-29; First posted 2024-05-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: GNAO1; Dystonia; Epilepsy; Development Delay; Developmental and Epileptic Encephalopathy 17; Neurodevelopmental Disorder With Involuntary Movements; Choreoathetosis
Keywords: GNAO1
MeSH Terms: conditions — Dystonia; Epilepsy; Learning Disabilities | interventions — Zinc Acetate

STUDY DESIGN:
Intervention Model Description: Prospective single arm, open-label pilot trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional Arm (Experimental): Zinc acetate dihydrate in age-adapted dosage ranging from 50mg to 150mg Zn2+ per day according to the recommended dosage in Wilsons Disease.
  Interventions: Drug: Zinc Acetate Dihydrate

INTERVENTIONS:
Drug: Zinc Acetate Dihydrate — In this single arm trial, all participants will be receive the trial drug zinc acetate dihydrate orally. The Investigational medicinal product (IMP) will be given one hour after meal in a dosage which is recommended in Wilson Disease and has been given in this condition without observing severe adverse effects. If oral administration is not possible due to the disability level of the patient, the IMP can be mortared and suspended and can then be given as suspension orally or via the Percutaneous endoscopic gastrostomy. The total treatment duration in each patient is 6 months with stable dosage over the duration of the trial. If the therapy shows effects, the parents and participants may continue medication after the end of the trial. If not, they will stop the medication after the last visit at the trial site.
  Other Names: WILZIN 25mg; WILZIN 50mg; Wilzin

SUMMARY:
The goal of this clinical trial is to investigate feasibility and safety of an oral therapy with zinc in patients affected by Guanine nucleotide-binding protein G(o) subunit alpha (GNAO1) associated disorders.

The main questions it aims to answer are:

* Is a daily oral therapy with zinc in GNAO1 associated disorders a safe and feasible therapy?
* Are there potential changes in general motor skills, general behaviour and well being, day/night rhythm, level of dyskinesia and dystonia, frequency of seizures, quality of life and changes in the microbiome of the patients.

Participants with GNAO1 associated disorders will be given an oral zinc therapy for 6 month and will be assessed in 3 visits and 2 phone calls within this trial.

ELIGIBILITY:
Inclusion Criteria:

* GNAO1 associated neurological disorder, documented by either

  * Proven pathogenic or likely pathogenic mutation in GNAO1 or
  * a variant of unknown significance in GNAO1 and clinical symptoms likely to be consistent with GNAO1 as determined by the investigators and
  * at least one of the common symptoms of GNAO1: Movement disorder (Dystonia, Chorea, Ataxia, clonic), central muscular hypotonia, epilepsy, global developmental delay
* Age: 6 month - 30 years
* GMFM ≤ 75
* written informed consent prior to any trial-related procedure (according to age and status of psycho-intellectual development)

  * of parents or legal guardian
  * of parents or legal guardian and patient
  * of the patient
* stable on following concomitant treatments for at least 3 months prior to trial inclusion: anti-seizure drugs (ASD); baclofen, Deep brain stimulation settings

Exclusion Criteria:

* Treatment of Zinc in the last 4 months before inclusion
* known other genetic variants that are known to cause symptoms like observed in GNAO1-related disorders, additional to the proven GNAO1 mutation
* implantation of Deep brain stimulation planned during the duration of the trial, i.e. in the six months after inclusion
* start of intrathecal baclofen therapy planned during the duration of the trial, i.e. in the six months after inclusion
* Known allergy/hypersensitivity to the scheduled trial drug
* Concomitant participation in other clinical drugs with investigational drugs or with competing interventions
* sexually active patients who are not willing to use/ not using a highly effective contraception method with a pearl-index < 1. Sexually active patients, unless surgically sterile, must be using a highly effective contraception method (including oral, transdermal, injectable or implanted contraceptives, intrauterine device (IUD), using a condom of the sexual partner or sterile sexual partner) and must agree to continue using such precautions during the whole study period.
* Pregnant women and nursing mothers

Ages: 6 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of daily treatment with oral zinc in GNAO1 as assessed by diary. | From first visit at Inclusion to visit after 6 month
  The feasibility is measured by the actual days that zinc was taken in the right dosage. If zinc was taken in the scheduled dosage at least on 80% of the days it is assumed to be feasible. Parents/caregivers document the daily intake into a diary.
Safety of daily administered zinc in GNAO1 as assessed by regular evaluation of the side effects | From first visit at inclusion until last phone call after 7 month
  To assess side effects: two phone calls are made and in each visit at site potential side effects are assessed.
Safety of daily administered zinc in GNAO1 as assessed by regular blood tests | Blood analysis at baseline, after 3 and 6 month
  Serum ferritin and copper detect potential deficiencies, caused by regular zinc administration and therefore reduced uptake. Liver enzymes, alkaline phosphates, lipase and amylase are assessed 3 times, since these parameters can be elevated as side effect.

SECONDARY OUTCOMES:
Level of motor-skills assessed by Gross-motor function measure | Compare measure at baseline to visit after 3 and 6 month
  The Gross-motor function measure(GMFM-66) is a standardized test for gross motor function, carried out by a physiotherapist. Minimum value 0, maximum value 100; a higher score is a better outcome.
Change in quality of life score assessed by Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) questionnaire for caregivers | Compare measure at baseline to visit after 3 and 6 month
  The CPCHILD questionnaire is a validated measure of health-related quality of life for children with severe disabilities and is evaluated 3 times in this trial. Parents/caregivers are asked to fill out the questionnaire. The CPCHILD currently consists of 37 items distributed among six sections representing the following domains:
  1. Activities of daily living/personal care (nine items)
  2. Positioning, transferring and mobility (eight items)
  3. Comfort and emotions (nine items)
  4. Communication and social interaction (seven items)
  5. Health (three items)
  6. Overall quality of life (one item) In Section 7, caregivers rate the importance of each of these items' contribution to their child's quality of life.Scores for each domain and for the total survey are standardized and range from a minimum: 0 (worse) to a maximum 100 (best). A higher score is a better outcome.
Level of Dystonia assessed by the Burke-Fahn-Marsden Dystonia Rating scale | Compare measure at baseline to visit after 3 and 6 month
  The Burke-Fahn-Marsden Dystonia Rating Scale is a universally applied instrument for the quantitative assessment of dystonia in both children and adults. It is divided into movement score and disability score. Movement score minimum value 0, maximum value 120; a higher score is a worse outcome with more dystonia present. Disability score minimum value 0; maximum value 30; a higher score is a worse outcome with more disabilities due to dystonia.
Level of dyskinesia assessed by the Abnormal involuntary movement scale (AIMS) | Compare measure at baseline to visit after 3 and 6 month
  The AIMS is a 12-item clinician-rated scale to assess severity of dyskinesias (specifically, orofacial movements and extremity and truncal movements) and will be assessed 3 times at each visit at site.
  The minimum score is 0 and the maximum score is 4 (severe). A higher score is a worse outcome showing higher level of dyskinesia.
Level of dyskinesia assessed by a movement log for parents/caregivers | Compare first two weeks of treatment to two weeks before the end of the trial
  Parents/caregivers are given a diary in which they are asked to document the hours per day which are disturbed by movement disorder and involuntary movements.
Changes in sleep assessed by diary for parents/caregivers | Compare first two weeks of treatment to two weeks before the end of the trial
  Parents/Caregivers are asked to fill out a diary addressing time of sleep per day and sleep disturbances.
Changes in general behaviour assessed by diary. | Compare answers of diary of first two weeks of treatment to two weeks before the end of the trial
  Parents/Caregivers are asked to fill out a diary addressing the general behaviour with two questions.
Changes in seizure frequency assessed by seizure log. | Compare first two weeks of treatment to two weeks before the end of the trial
  Parents/Caregivers are requested to document frequency in a seizure log which is part of the diary
Changes in seizure duration assessed by seizure log. | Compare first two weeks of treatment to two weeks before the end of the trial
  Parents/Caregivers are requested to document duration of seizures in a seizure log which is part of the diary
Changes in serum level of zinc assessed by regular blood analysis | Serum controls at baseline, after 3 and 6 month
  Serum controls of zinc are assessed three times to measure the changes in serum levels of zinc before and while zinc administration
Microbiome of stool assessed by regular analysis | Samples compared from baseline to samples collected after 3 and 6 month
  Analyze of the microbiome in stool to detect changes under therapy with oral zinc.The stool samples should be collected at home in the three days before visit 2 and 3 in special sample tubes that are handed out to the patient at visit 0. The first stool samples should be collected at visit 0 or on the first three days thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Thiel, MD, Principal Investigator — Children's Hospital, University Hospital Cologne, University of Cologne
Locations (1):
- Children's Hospital, University Hospital Cologne, University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No
Trial results will be published in a scientific journal and presented at national or international congresses. Publication of the results of the trial as a whole is intended. Anonymized individual patient data (IPD) can be made available on reasonable request to the PI after the results are published.

REFERENCES:
- [Background] Larasati YA, Savitsky M, Koval A, Solis GP, Valnohova J, Katanaev VL. Restoration of the GTPase activity and cellular interactions of Galphao mutants by Zn2+ in GNAO1 encephalopathy models. Sci Adv. 2022 Oct 7;8(40):eabn9350. doi: 10.1126/sciadv.abn9350. Epub 2022 Oct 7. PMID 36206333
- [Background] Thiel M, Bamborschke D, Janzarik WG, Assmann B, Zittel S, Patzer S, Auhuber A, Opp J, Matzker E, Bevot A, Seeger J, van Baalen A, Stuve B, Brockmann K, Cirak S, Koy A. Genotype-phenotype correlation and treatment effects in young patients with GNAO1-associated disorders. J Neurol Neurosurg Psychiatry. 2023 Oct;94(10):806-815. doi: 10.1136/jnnp-2022-330261. Epub 2023 May 24. PMID 37225406
- [Background] Briere L, Thiel M, Sweetser DA, Koy A, Axeen E. GNAO1-Related Disorder. 2023 Nov 9. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK597155/ PMID 37956232
- [Background] Savitsky M, Solis GP, Kryuchkov M, Katanaev VL. Humanization of Drosophila Galphao to Model GNAO1 Paediatric Encephalopathies. Biomedicines. 2020 Oct 6;8(10):395. doi: 10.3390/biomedicines8100395. PMID 33036271
- [Derived] Larasati YA, Solis GP, Koval A, Korff C, Katanaev VL. A Personalized 14-3-3 Disease-Targeting Workflow Yields Repositioning Drug Candidates. Cells. 2025 Apr 8;14(8):559. doi: 10.3390/cells14080559. PMID 40277885